CLINICAL TRIAL: NCT05803564
Title: Clinical Application of a New Technique of Thoracoabdominal Aortic Stent System for Endovascular Treatment of Thoracoabdominal Aortic Dissecting Aneurysm.
Brief Title: Thoracoabdominal Aortic Stent System for Endovascular Treatment of Thoracoabdominal Aortic Dissecting Aneurysm.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guard-FIM-01
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Thoracoabdominal; Aortic, Aneurysm, Dissecting
Keywords: Thoracoabdominal aortic stent system; thoracoabdominal aortic dissecting aneurysm; G-Branch
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Endovascular treatment of patients withThoracoabdominal Aortic Aneurysm using multibranched stent graft system
  Interventions: Device: Thoracoabdominal aortic stent system

INTERVENTIONS:
Device: Thoracoabdominal aortic stent system — Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with thoracoabdominal aortic stent system.

SUMMARY:
A First in man study to evaluate the safety and efficacy of thoracoabdominal aortic stent system for endovascular treatment of thoracoabdominal aortic dissecting aneurysm.

DETAILED DESCRIPTION:
The study is mainly for patients with thoraco-abdominal aortic dissecting aneurysm, and all subjects who passed the screening and signed the informed consent will be enrolled. Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with thoracoabdominal aortic stent system. Patients will be followed up at discharge, 1 month, 6 months, 12 months after the implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged greater than 18 years old and less than 80 years old;
2. Patients diagnosed with thoraco-abdominal aortic dissecting aneurysm and at least one of the following conditions should be met:

   a)Maximum aneurysm diameter >50 mm; b）Increase in diameter by more than 5 mm in recent 6 months c）Symptoms such as abdominal pain and back pain associated with thoracic and abdominal aortic dissecting aneurysm were identified.

   d）Poor morphology of thoracic and abdominal aortic dissecting aneurysm; e）Aortic dissection tears to iliac artery resulting in common iliac artery dissection tumor diameter >40 mm;
3. Anatomic criteria

   a)The diameter of the proximal anchoring area (aorta or implanted graft) ranged from 17~36 mm to ≥25 mm in length; b）Distal anchoring area (aorta or implanted graft): If distal anchoring area is in iliac artery, anchoring area diameter range 7~25 mm, length ≥15 mm; If the distal anchoring area is in the abdominal aorta, the anchoring area has a diameter of 12~36 mm and a length of ≥20 mm; c）There is a normal anchoring area at the distal end of the visceral branch vessel. The diameter range of the anchoring area is 6~13 mm and the length is ≥15 mm.

   d）Normal anchoring zone at distal renal artery, anchoring zone diameter 4.5~9 mm, length ≥15 mm; e）Suitable iliac, femoral, and upper limb arterial access.
4. Patients who understand the purpose of the trial, volunteer to participate and sign the informed consent form, and are willing to complete follow-up as required by the protocol;

Exclusion Criteria:

1. Patients with severe hematoma in aortic wall in proximal anchoring area of stent
2. Patients requiring simultaneous coverage and embolization of bilateral internal iliac arteries;
3. Patients with a history of acute coronary syndrome within 6 months; Acute coronary syndromes are cardiac acute ischemic syndromes resulting from rupture of an unstable atherosclerotic plaque in the coronary artery or erosion secondary to the formation of new blood 4 thrombus, including ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, and unstable angina.
4. Patients with a transient ischemic attack (TIA) or ischemic/hemorrhagic stroke within 3 months;
5. Patients with preoperative hepatic and renal dysfunction [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the normal upper limit; Serum creatinine (Cr) >150u mol/L];
6. Patients with severe pulmonary insufficiency who cannot tolerate general anesthesia;
7. Patients with severe coagulopathy;
8. Patients with a history of hypersensitivity to contrast agents, anticoagulants, antiplatelet agents, stent delivery devices (i.e., nitinol, polyester, PTFE, nylon polymer materials);
9. Patients with connective tissue diseases such as systemic lupus erythematosus, Marfan syndrome, Egyptian syndrome, or Behcet's disease;
10. Patients with arteritis;
11. Patients with significant organ dysfunction or other serious disease;
12. Women with planned pregnancy, pregnancy stage , or lactation;
13. The patient participated in another clinical trial and was not out or withdrawn within the first 3 months of the screening period of this trial.
14. Patients with a life expectancy of not more than 1 year;
15. Patients judged by the investigator to be unsuitable for endovascular treatment;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Major Adverse Events (MAE) Within 30 Days Postoperative | within 30 days postoperative
  Major Adverse events (MAE) are defined as death related to thoracic and abdominal aortic dissecting aneurysms, stroke, permanent paraplegia, kidney failure, intestinal necrosis, myocardial infarction, respiratory failure, and liver failure.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Professor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No